CLINICAL TRIAL: NCT00321815
Title: A Randomized Phase 2 Trial Of Erlotinib With Or Without PF-3512676 For The Treatment Of Patients With Advanced EGFR-Positive Non-Small Cell Lung Cancer After Failure Of At Least One Prior Chemotherapy Regimen
Brief Title: Trial Of Erlotinib With Or Without PF-3512676 In Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8501006
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: advanced carcinoma non-small cell lung EGFR positive Erlotinib Tarceva PF-3512676 Phase II immunotherapy immune modulator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ProMune; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Standard of Care chemotherapy plus experimental intervention (PF-3512676)
  Interventions: Drug: PF-3512676 + Erlotinib
- B (Active Comparator): Standard of Care chemotherapy
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: PF-3512676 + Erlotinib — PF-3512676 0.2 mg/kg subcutaneously on days 1, 8 and 15 of each 21 day cycle until disease progression or unacceptable toxicity.
  Erlotinib 150 mg orally daily (21 day cycles) until disease progression or unacceptable toxicity
  Arms: A
Drug: Erlotinib — Erlotinib 150 mg orally daily (21 day cycles) until disease progression or unacceptable toxicity
  Other Names: Tarceva
  Arms: B

SUMMARY:
To assess the efficacy and safety of PF-3512676 administered in combination with erlotinib in patients with advanced EGFR-positive non-small cell lung cancer after failure of at least one prior chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, EGFR-positive NSCLC
* ECOG Performance Status 0, 1 or 2
* Measurable disease

Exclusion Criteria:

* Known CNS metastasis
* Pre-existing autoimmune or antibody mediated disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 50Events

SECONDARY OUTCOMES:
Overall Safety Profile | 28 days post treatment
Time to Tumor Progression | End of treatment
Overall Objective Response Rate | Time of disease progression
Duration of Response | Time of disease progression
Overall Survival | Time of death

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - Pfizer Investigational Site, Daphne, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Corona, California
  - Pfizer Investigational Site, Glendora, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Pomona, California
  - Pfizer Investigational Site, Rancho Cucamonga, California
  - Pfizer Investigational Site, San Mateo, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Deerfield Beach, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Mason City, Iowa
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Bridgeton, Missouri
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Kirkwood, Missouri
  - Pfizer Investigational Site, Somerville, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Fairfield, Ohio
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Philadephia, Pennsylvania
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Dalls, Texas

REFERENCES:
- [Derived] Belani CP, Nemunaitis JJ, Chachoua A, Eisenberg PD, Raez LE, Cuevas JD, Mather CB, Benner RJ, Meech SJ. Phase 2 trial of erlotinib with or without PF-3512676 (CPG 7909, a Toll-like receptor 9 agonist) in patients with advanced recurrent EGFR-positive non-small cell lung cancer. Cancer Biol Ther. 2013 Jul;14(7):557-63. doi: 10.4161/cbt.24598. Epub 2013 May 10. PMID 23792641
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8501006&StudyName=Trial%20Of%20Erlotinib%20With%20Or%20Without%20PF-3512676%20In%20%20Advanced%20Non%20Small%20Cell%20Lung%20Cancer%0A